CLINICAL TRIAL: NCT01266785
Title: Analysis of Relationship Between Infliximab Treatment Response, Regulatory T Cells, and Interleukin-2 in Crohn's Disease
Brief Title: Infliximab, Regulatory T Cells, IL2 and Crohn's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Judy Collins, Physician, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6572
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Crohn's Disease
Keywords: crohn's; Infliximab; Inflammatory bowel disease; digestive tract; Interleukin
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Infliximab — Patient will receive Infliximab infusions during Weeks 0, 2 and 6. Therefore, the duration of the Infliximab treatment will last 6 weeks.

SUMMARY:
Crohn's disease is an inflammatory (swelling and soreness) disorder of the digestive tract. Affected patients suffer from abdominal pains, diarrhea (sometimes bloody), weight loss. It is a lifelong disease with frequent flares during the course of the disease. Crohn's disease is mostly treated with medications, sometimes surgery is needed. Infliximab is a medication for treating severe Crohn's disease. This medicine is effective by blocking special substance (tumor necrosis factor) released from certain white blood cells in the body. Infliximab is given via a vessel at week 0, 2, 6 initially, then every 2 monthly for maintenance. However, some of patients with Crohn's disease do not respond infliximab. Currently there is no test to reveal which patients will respond to treatment. This study aims to analyze and compare particular subgroup of white cells and its products during and after infliximab treatment which may determine the responsiveness to infliximab treatment.

DETAILED DESCRIPTION:
All patients will have chest x-ray and pregnancy test (if female) prior to infliximab treatment.

There will be total 5 study visits. At each visit, body weight will be measured, abdominal exam will be performed , 2 tablespoonful of blood will be drawn, stool will be collected, a questionnaire will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or exacerbating CD (Moderate to severe CD).
* The diagnosis of moderate to severe CD will be confirmed by previous endoscopy and biopsy.
* Have the capacity to understand and sign an informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Changes of IL-2 and Treg cell levels | 1 year
  To determine if the change of IL-2 and Treg cell levels can be used clinically as a predictive marker for differentiating Infliximab responders from nonresponders

CONTACTS AND LOCATIONS:
Overall Officials: Zili Zhange, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Boschetti G, Nancey S, Sardi F, Roblin X, Flourie B, Kaiserlian D. Therapy with anti-TNFalpha antibody enhances number and function of Foxp3(+) regulatory T cells in inflammatory bowel diseases. Inflamm Bowel Dis. 2011 Jan;17(1):160-70. doi: 10.1002/ibd.21308. PMID 20848510
- [Background] Di Sabatino A, Biancheri P, Piconese S, Rosado MM, Ardizzone S, Rovedatti L, Ubezio C, Massari A, Sampietro GM, Foschi D, Porro GB, Colombo MP, Carsetti R, MacDonald TT, Corazza GR. Peripheral regulatory T cells and serum transforming growth factor-beta: relationship with clinical response to infliximab in Crohn's disease. Inflamm Bowel Dis. 2010 Nov;16(11):1891-7. doi: 10.1002/ibd.21271. PMID 20848485
- [Background] Li Z, Arijs I, De Hertogh G, Vermeire S, Noman M, Bullens D, Coorevits L, Sagaert X, Schuit F, Rutgeerts P, Ceuppens JL, Van Assche G. Reciprocal changes of Foxp3 expression in blood and intestinal mucosa in IBD patients responding to infliximab. Inflamm Bowel Dis. 2010 Aug;16(8):1299-310. doi: 10.1002/ibd.21229. PMID 20196149
- [Background] Ricciardelli I, Lindley KJ, Londei M, Quaratino S. Anti tumour necrosis-alpha therapy increases the number of FOXP3 regulatory T cells in children affected by Crohn's disease. Immunology. 2008 Oct;125(2):178-83. doi: 10.1111/j.1365-2567.2008.02839.x. Epub 2008 Apr 16. PMID 18422560